CLINICAL TRIAL: NCT04242511
Title: Comparison of Anti-tuberculous Drug Levels in Diabetic and Non-diabetic Tuberculosis Patients
Brief Title: Tuberculosis Drug Levels in Diabetics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: v1.0 30/10/2019
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Tuberculosis; Diabetes Mellitus
Keywords: Tuberculosis; Diabetes; Rifampicin; Therapeutic Drug Monitoring
MeSH Terms: conditions — Tuberculosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Blood samples will be taken and analysed by high performance liquid chromatograp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Tuberculosis patients with diabetes mellitus:
  1. Subject aged 18 years of age or over
  2. Written, informed consent obtained.
  3. New diagnosis of tuberculosis and started on anti-tuberculosis treatment
  4. Known diagnosis of diabetes or two consecutive raised IFCC HbA1c levels (>= 48 mmol/mol) at the time of TB diagnosis
  Interventions: Diagnostic Test: Measurement of tuberculosis medications level
- Controls: Tuberculosis patients without diabetes mellitus:
  1), 2), 3) as above 4) IFCC HbA1c level < 48mmol/mol 5) Weight matched to cases (+/- 2kg)
  Interventions: Diagnostic Test: Measurement of tuberculosis medications level

INTERVENTIONS:
Diagnostic Test: Measurement of tuberculosis medications level — Measurement of tuberculosis medication levels at 2 hours post-dose

SUMMARY:
This study compares blood levels of tuberculosis medications between diabetic patients and non-diabetic patients. There is some research that suggests these medications are at lower levels in diabetic patients with tuberculosis, and this could adversely affect the outcome of their infection. Diabetic patients are at higher risk of dying or having a severe episode of tuberculosis therefore it is important that their care is optimised as far as possible.

To answer the research question all participants in the study will have an extra blood sample drawn at the same time as their routine blood tests which are used to monitor their tuberculosis treatment. Some participants will have additional blood samples taken at different times to give a more accurate picture of the medication levels in their bloodstream. The study will be conducted in the tuberculosis clinics at London North West University Healthcare NHS Trust and will include adult patients with and without diabetes who have recently been diagnosed with tuberculosis.

Some other information about their routine medications, weight and height, and severity of diabetes will also be collected, to see if these affect the medication levels in the bloodstream as well.

DETAILED DESCRIPTION:
This is a case-controlled study measuring tuberculosis medication levels in diabetic and non-diabetic patients on treatment for tuberculosis.

Case:

Our tuberculosis clinic checks the levels of glycosalated haemoglobin (HbA1c), a marker of diabetes, in all patients with a new diagnosis of tuberculosis before they start treatment. All patients who are either known to have diabetes or have a raised HbA1c level will be identified at their clinic appointment. Patients who have a raised HbA1c and are not known to have diabetes will have a repeat blood test to confirm the result as part of normal clinical practice. If their level is still raised or they are known to have diabetes they will be asked if they wish to participate in the study.

They will be provided with a patient information leaflet and given the opportunity to ask questions, and discuss with friends and family if preferred.

If they agree to participate their tuberculosis care will continue as usual. Part of the standard care for our TB patients is to have blood tests at 2 weeks, 4 weeks and 8 weeks after starting treatment, to check for toxicity from the medications.

They will be asked to take their TB medications as usual on the morning of their scheduled blood tests.

To confirm the time at which they took their doses they will be asked to either take a time-stamped video of themselves taking their morning tablets, or to text or call the study co-ordinator when they take their tablets. They will then be asked to come in for the blood test 2 hours later. Prior to the blood test their consent will be confirmed and they will be given the opportunity to ask questions or withdraw from the study. Along with the routine blood tests (to check full blood count, liver and kidney functions) a further sample will be taken to check levels of the TB medications.

They will also have their weight checked, and be asked if their other medications (eg for diabetes) have changed since their first clinic appointment.

If they are known to have abdominal tuberculosis, or are suspected to have other problems with absorbing food and medications, they will be asked to stay for a second blood test between 0 and 8 hours after they took their medication. This will help identify the peak medication level more accurately if absorption from the gut is delayed.

A small number of the diabetic patients may also be asked to inform the study co-ordinator when they take their anti-diabetic medications so that the study blood sample can also be used to measure the levels of their anti-diabetic medications.

The blood samples for the routine tests will be processed by the hospital pathology lab as usual. Study blood samples will be spun to separate the serum which contains the medications. The serum will then be frozen at -20C, prior to being processed in batches using High Performance Liquid Chromatography.

If the participant agrees the same procedure will be carried out at their 4 and 8 week routine blood tests.

Controls:

Controls will be recruited from TB clinic in a similar way to cases. Patients who have an HbA1c level <48 mmol/mol and no history of diabetes will be reviewed to see if they meet the eligibility criteria. This will include assessing whether they are in the same weight category (5kg bands e.g. 50-54kg, 55-59kg, 60-64kg etc) as recruited diabetic patients. If they consent to participate then they will be asked to follow the same study protocol as the diabetic cases, as detailed above.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 18 years of age or over
2. Written, informed consent obtained.
3. New diagnosis of tuberculosis and started on anti-tuberculosis treatment Cases: Known diagnosis of diabetes or two consecutive raised IFCC HbA1c levels (>= 48 mmol/mol) at the time of TB diagnosis Controls: IFCC HbA1c level < 48mmol/mol

Exclusion Criteria:

1. Subject aged under 18 years
2. Inability to give informed consent
3. Repeat HbA1c level <48mmol/mol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in the tuberculosis clinics at London North West University Healthcare NHS Trust. The study participants will be recruited from patients with a diagnosis of tuberculosis, with and without diabetes. Diabetes is a common comorbidity in tuberculosis patients in this area, with a prevalence of around 15 to 20%.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
TB medication levels | 2 hours following medication dose
  Comparison of 2-hour post-dose levels of anti-tuberculosis medications

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Barrett, Principal Investigator — LONDON NORTH WEST UNIVERSITY HEALTHCARE NHS TRUST

IPD SHARING:
Plan to Share IPD: Undecided